CLINICAL TRIAL: NCT04627805
Title: Reproductive Decision Support Tool for Women With Substance Use Disorders: A Pilot Study
Brief Title: Evaluating MyPath to Enhance Reproductive Autonomy and Liberate Decision-making
Acronym: EMERALD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment hindered by COVID-19 pandemic, unable to recruit participants virtually
Sponsor: University of Pittsburgh (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Principal Investigator, Beatrice Chen, Associate Professor, University of Pittsburgh
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY20010128
Record Dates: First submitted 2020-11-08; First posted 2020-11-13 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Substance Use Disorders; Reproductive Issues; Contraception
Keywords: Reproductive decisions; Pregnancy planning; Contraceptive counseling
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: The investigators will enroll the first 33 participants to the usual care group, to evaluate the baseline occurrence of family planning discussions and referrals. Following the completion of the usual care group, the investigators will then enroll 33 participants to the MyPath intervention. This allocation scheme was chosen so as to not contaminate the baseline group by rolling out the intervention simultaneously.
  Providers will be recruited at the conclusion of the study to complete an exit survey if they interacted with at least one Phase 3 participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 2: Usual Care (No Intervention): The investigators will enroll 33 women with SUDs to evaluate baseline family planning discussions and referrals to women's health providers in SUD treatment settings. To establish usual care practice patterns, MyPath will not be administered to this group of participants. Participants will be asked to complete a pre-visit survey, including substance use history and current reproductive health goals, as well as questions about reproductive health knowledge, self-efficacy, and decision conflict. The participants will then attend their scheduled therapy visit with the substance use treatment provider. Following the therapy visit, they will complete the post-visit survey, which will include the same knowledge, efficacy, and decision conflict survey questions as the pre-visit survey. Occurrence of reproductive health discussions, prescriptions or referrals, and satisfaction with reproductive health services will be measured following the visit as well.
- Phase 3: MyPath Pilot (Experimental): Following completion of the usual care arm, the investogators will enroll a second group of 33 women with SUDs to participate in the MyPath intervention arm. Participants will complete the same pre-visit survey as the usual care group. In addition, they will be provided a website link to navigate through the online MyPath tool. Following completion of MyPath, participants will receive a summary page that they will be encouraged to use as a guide when discussing their reproductive health with their substance use treatment provider at their next scheduled therapy visit. After the visit, they will complete the post-visit survey. In addition to satisfaction with reproductive health services, the intervention group will be asked specific questions about their perception of the MyPath tool.
  Interventions: Behavioral: MyPath tool

INTERVENTIONS:
Behavioral: MyPath tool — MyPath is a reproductive decision support tool that utilizes a patient-centered approach to help women frame their reproductive decisions in the context of their goals, preferences, and health needs. This tool was developed by Dr. Lisa Callegari with funding from the Veterans Administration (VA) Health Services Research & Development to be used in primary care settings with women veterans. It is conceptually grounded in Self-Determination Theory, which postulates that health care that meets patients' psychological needs in three key domains - autonomy, competence, and relatedness - will result in improved health behaviors and health outcomes. This is particularly relevant in reproductive health care, given the highly individualized and personal nature of these decisions, and the importance of centering a woman's aspirations and goals in her health care decision making.
  Arms: Phase 3: MyPath Pilot

SUMMARY:
This is a pilot study to evaluate the acceptability and feasibility of incorporating a patient-facing reproductive decision support tool, MyPath, into existing clinical pathways in a SUD treatment program. This study will be conducted virtually in partnership with a single substance use treatment program within the University of Pittsburgh Medical Center (UPMC).

Aim 1: Assess the feasibility and acceptability of incorporating a patient-facing reproductive decision support tool (MyPath) into existing clinical pathways in a substance use treatment program.

Aim 2: Assess preliminary efficacy of MyPath on reproductive health knowledge, self-efficacy, and decisional conflict as compared to usual care, as well comparisons between receipt of reproductive health services during the usual care period versus after implementing the intervention.

The investigators hypothesize that the MyPath tool is acceptable and feasible for participants and their providers within a SUD treatment program. They also anticipate that preliminary efficacy data will show a positive correlation between the MyPath intervention and receipt of reproductive services, as well as increased knowledge and self-efficacy with decreased decision conflict. This pilot study will lay the groundwork for future larger trials in order to measure efficacy of this tool in substance use treatment settings.

DETAILED DESCRIPTION:
The study will be completed in four phases.

Phase 1 (Preparation): First, a sample of women with SUDs (n=5) will be recruited through a separate MAT program in the UPMC system to pre-test the surveys for patient participants to ensure clarity and understandability of these assessments. A sample of substance use treatment providers (n=3) will also be recruited to pre-test the surveys for provider participants. To ensure that participants who want contraceptive services can receive them, the investigators will create a referral pathway that can be used to link participants interested in receiving reproductive health services to an appropriate provider. Through the electronic medical record system of UPMC, providers at NATP will be able to place referrals for reproductive health services for interested participants. Additionally, given the recent increase in use of telemedicine during the COVID-19 pandemic, participants will have the option of attending a telemedicine video visit with a family planning provider through UPMC Magee-Womens Hospital's Family Planning clinic. These various options will allow participants to choose the route that is easiest for them and therefore will further decrease barriers to care.

Phase 2 (Usual Care): Thirty three women with SUDs will be recruited from the NATP to evaluate baseline family planning discussions and referrals to women's health providers in SUD treatment settings. To establish usual care practice patterns, MyPath will not be administered to this group of participants. Participants will first complete a pre-visit survey. This will include demographics, substance use history, and current reproductive health goals, as well as questions about knowledge, self-efficacy, and decision conflict. The participants will then attend their scheduled visit with the substance use treatment provider, whether virtual or in-person. Following the provider visit, they will complete the post-visit survey, which will include the same knowledge, efficacy, and decision conflict survey questions as the pre-visit survey. Occurrence of reproductive health discussions, prescriptions or referrals, and satisfaction with reproductive health services will be measured following the visit as well. All surveys will be administered online through REDCap. Patient participants will be compensated for their time with a gift card after they complete the post-visit survey.

Phase 3 (MyPath Pilot): Following completion of the usual care arm, a second group of 33 women with SUDs will be recruited from the NATP to participate in the MyPath intervention arm. Participants will complete the same pre-visit survey as the usual care group. In addition, they will be provided a website link to navigate through the online MyPath tool. Following completion of MyPath, participants will receive a summary page (see Appendix A for a sample summary) that they will be encouraged to share with their substance use treatment provider at their next scheduled visit, whether virtual or in-person. After the visit, they will complete the post-visit survey. In addition to satisfaction with reproductive health services, the intervention group will be asked specific questions about their perception of the MyPath tool. All surveys will be administered online through REDCap. Patient participants will be compensated for their time with a gift card after they complete the post-visit survey.

Phase 4 (Provider Assessment): Following study completion for patient participants, provider participants will be asked to complete an exit survey to assess feasibility of incorporating MyPath into their clinical work flow and their comfort with reproductive counseling and referring. This will be an anonymous survey administered online and will be sent to all providers identified as engaging with at least one patient participant during the MyPath intervention.

Phase 5 (Follow-up): Three months following study completion, a chart review will be performed for each patient participant through UPMC's electronic medical record. This will allow for the collection of information for completion of placed referrals and receipt of desired reproductive services.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged 18-45 years
* Enrolled in a substance use treatment program
* English-speaking
* Interested in discussing their reproductive health with their substance use provider
* Willing and able to participate in a virtual study using video and/or phone

Exclusion Criteria:

* Currently pregnant
* History of female sterilization, hysterectomy, bilateral oophorectomy, or monogamous with a partner with vasectomy
* Previously enrolled in the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Number of participants reporting satisfaction with reproductive discussions assessed by 5-point Likert scale | Approximately 2 weeks
  Number of participants that report they are somewhat satisfied or very satisfied with reproductive discussions as assessed on a Likert scale from 1 (very dissatisfied) to 5 (very satisfied)
Number of providers reporting comfort with reproductive discussions assessed by 5-point Likert scale | Approximately one month
  Number of providers that report they are comfortable or very comfortable with reproductive discussions as assessed on a Likert scale from 1 (very uncomfortable) to 5 (very comfortable)
Number of participants reporting satisfaction with MyPath assessed by 5-point Likert scale | Approximately 2 weeks
  Number of participants that report they agree or strongly agree with satisfaction statements about MyPath as assessed on a Likert scale from 1 (strongly disagree) to 5 (strongly agree)
Number of providers reporting satisfaction with MyPath assessed by 5-point Likert scale | Approximately one month
  Number of providers that report they agree or strongly agree with satisfaction statements about MyPath as assessed on a Likert scale from 1 (strongly disagree) to 5 (strongly agree)

SECONDARY OUTCOMES:
Number of providers reporting ease of incorporating MyPath into clinical workflow assessed by 5-point Likert scale | Approximately one month
  Likert scale Number of providers that report they agree or strongly agree with ease of incorporation statements about MyPath as assessed on a Likert scale from 1 (strongly disagree) to 5 (strongly agree)
Number of participants who complete all study procedures | Approximately six months
  Number of participants who enroll and complete all study procedures, including enrollment visit, pre- and post-surveys, and MyPath tool
Mean change in reproductive health knowledge | Approximately one month
  Mean change in reproductive health knowledge defined as the difference in the number of correct responses to a set of reproductive health knowledge questions from surveys administered before and after the study visit
Mean change in self-efficacy | Approximately one month
  Mean change in self-efficacy, as assessed on a 5-point Likert scale from 1 (not confident at all) to 5 (very confident) by a set of self-efficacy statements from surveys administered before and after the study visit
Mean change in decisional conflict | Approximately one month
  Mean change in decisional conflict, as assessed on a 5-point Likert scale from 1 (strongly disagree) to 5 (strongly agree) by a set of decision statements from surveys administered before and after the study visit
Number of participants who received reproductive health services | Approximately four months
  Number of participants who received reproductive health services as assessed by medical chart review at three month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice A Chen, MD MPH, Principal Investigator — University of Pittsburgh; Samantha J Deans, MD MPH, Study Director — University of Pittsburgh
Locations (1):
- Center for Family Planning Research, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Teal S, Haider S, Harris L, Hubacher D, Raine-Bennett T. Scientific abstracts: Featured research at the 2019 Society of Family Planning Annual Meeting. Contraception. 2019 Jul 23:303-304. doi: 10.1016/j.contraception.2019.07.007. Online ahead of print. No abstract available. PMID 31472941
- See also: MyPath web-based decision support tool — http://www.mypathtool.org